CLINICAL TRIAL: NCT01599975
Title: Phase III, Placebo-Controlled, Double-Blind Crossover Study of Slow-Release Methylphenidate (Concerta ™) for Treatment of HIV Associated Neurocognitive Disorder
Brief Title: A Study Comparing Long-acting Methylphenidate (ConcertaTM) vs. Placebo in the Treatment of Memory Loss Due to HIV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ardis Ann Moe, M.D., Associate Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Concerta HIV Study
Record Dates: First submitted 2012-05-07; First posted 2012-05-16 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: HIV Dementia
Keywords: HAND; HIV Associated Neurocognitive Disorder; Methylphenidate; HIV Dementia
MeSH Terms: conditions — AIDS Dementia Complex | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A: 2 tabs of 18 mg Concerta daily (Active Comparator): 20 subjects to receive active study drug in a blinded fashion x 2 weeks, then washout x 2 weeks, then cross over to receive matched placebo x 2 weeks.
  Interventions: Drug: Long acting methylphenidate
- Group B: Matched placebo, 2 tabs daily (Placebo Comparator): Group B to receive matched placebo x 2 weeks, then washout x 2 weeks, then cross over to receive active drug in a blinded fashion x 2 weeks.
  Interventions: Drug: Matched placebo

INTERVENTIONS:
Drug: Long acting methylphenidate — Treatment with long-acting methylphenidate, 36 mg a day as 2 tablets of 18 mg each.
  Other Names: Concerta
  Arms: Group A: 2 tabs of 18 mg Concerta daily
Drug: Long acting methylphenidate — 18 mg tablets, 2 tablets daily by mouth x 2 weeks, then washout x 2 weeks, then crossover to 2 tablets of matched placebo x 2 weeks.
  Arms: Group A: 2 tabs of 18 mg Concerta daily
Drug: Matched placebo — 2 tablets of matched placebo daily by mouth
  Other Names: Matched placebo as supplied by Johnson and Johnson
  Arms: Group B: Matched placebo, 2 tabs daily

SUMMARY:
This study is being done to see if a drug called long acting methylphenidate (Concerta) is safe and effective as a treatment for problems with mental function in adults infected with HIV.

A subset of patients with HIV-associated memory loss have a defect in the speed with which they learn and process information. Methylphenidate drugs, such as Ritalin or Concerta, have been shown on tests to improve the ability to rapidly absorb information; these tests are called "reaction time tests". These drugs are already FDA-approved to treat Attention Deficit Disorders: ADD or ADHD.

At baseline, all subjects get tests of memory and brain function; then they are split into two groups. One group on this study will receive Concerta for 2 weeks, and a second group will receive a placebo x 2 weeks. After that period both groups will receive memory and other tests of brain function, and then the groups will switch. The first group will receive placebo and the second will receive Concerta x 2 weeks, followed by more memory and neurological tests. After that all subjects will have the option to receive Concerta for free for 8 more weeks. At the last visit all subjects get memory and brain tests again.

DETAILED DESCRIPTION:
There are 11 study visits in 14 weeks.

In Part I of the study one-half of the subjects will receive ConcertaTM and one-half will receive placebo.

After 2 weeks all subjects will stop their study medication for 2 week (the "washout period"), and then all of the subjects who received placebo will then receive 2 weeks of methylphenidate, and all of the subjects who received long acting methylphenidate will receive placebo for 2 weeks.

The subject will be invited to enter Part II of the study if she/he still qualifies. During this portion of the study, the subject will receive ConcertaTM for 8 weeks. The subject does not have to be on Part II of this study to be on this study.

Screening visit. (4 hours)

There is a screening medical visit. If the subject passes the initial questions for depression and dementia, the subject will undergo the following procedures:

There will be a physical examination including a medical and medication history, which will include telling the study staff about all of the drugs that the subject has taken recently or are currently taking, and measurement of vital signs (blood pressure, temperature, height, weight, pulse,breathing rate).

The subject will have a physical examination including a detailed test of reflexes, muscle strength,gait, balance, and other functions of brain and nerves to see if he/she has any nerve damage and to see how the brain functions. The subject will take a group of tests called neuropsychological tests. The subject will answer questions, do simple tasks with their hands, and see how long it takes her/him to walk a short distance. Some of these questions are to test the subject for depression and memory abilities.

The subject will need to bring in your most recent CD4 cell count (T-cell counts) and HIV viral load on this visit.

If the initial screening questionnaires show that the subject fulfills some of the requirements of the study, the subject will be asked to have about 2 tablespoons of blood drawn from a vein in his/her arm, a urine test for drugs of abuse, and a urine pregnancy test if the subject is female and able to bear children. Some of the blood tests are to measure liver and kidney function and to see if the subject is anemic. The subject will have an EKG (electrocardiogram).

. Entry Visit (Week 0) If the subject qualifies for this study the subject will return to the clinic for an entry visit. The entry visit will occur within 2 weeks of Visit 1. This visit will take about 3-4 hours. At this visit you will undergo the following procedures: The subject will have a short physical examination and be asked questions about your health and the medications she/he is taking. The subject will be asked to complete another set of tests of memory and mental function. If the subject is a woman of child bearing potential he/she will have a pregnancy test at this visit and every 4 weeks thereafter. Once the subject has completes the entry tests, she/he will be assigned by chance (like flipping a coin) to either ConcertaTM, or placebo.

The study treatment groups are:

Group A: ConcertaTM 2 tablets taken with food in the morning OR Group B: Placebo, 2 tablets taken with food in the morning.

The first dose of study medication will be given in the clinic. She/he will be asked to take 1 tablet of study medication in the clinic and be observed for 2 hours afterward to see if you have any immediate side effects. The blood pressure will be checked again. The first dose of study medication is only 1 tablet of the study medication. On the day after this clinic visit she/he will take your second dose of study medication. This will be 2 tablets of study medication. Thereafter the subject will be taking 2 tablets of study medication in the morning. The study medications will be given as a 2-week supply.

Week 1 Visit (1 hour) The subject will be asked brief medical questions and receive a brief physical exam with vital signs and an EKG if indicated. She/he will be asked for a urine sample. She/he will have one short memory test.

Week 2 Visit (3 hours) He/she will be asked to come to clinic before he/she takes the daily dose of study medication. He/she are asked to bring your study medications with them, and to take the study medication in the presence of the study staff, who will note the time. He/she will be asked brief medical questions and receive a brief physical exam and a detailed test of his/her brain and nerve function. He/she will have an EKG and a blood test of about 2 tablespoons to check liver and kidney function, and to check for anemia.

She/he will also be asked questions about emotions, memory function, and ability to do simple tasks. If she is a woman able to become pregnant she will be asked to have a urine pregnancy test. After this visit the subject will stop taking study medications for 2 weeks (2 week washout period).

Week 4 (4 hours) He/she will be asked brief medical questions and receive a brief physical exam, and a detailed test of brain and nerve function. He/she will be asked questions about emotions, memory function, and ability to do simple tasks. He/she will be given a new supply of study medications. The subject will be asked to take 1 tablet of study medication in the clinic and be observed for 2 hours afterward to see if he/she has immediate side effects. Blood pressure will be checked again. On the day after this clinic visit the subject will take 2 tablets of study medication. Thereafter the subject will be taking 2 tablets of study medication in the morning.

Week 5 (1 hour) The subject will be asked brief medical questions and receive a brief physical exam and an EKG if indicated. The subject will be asked for a urine sample. He/she will have one short memory test.

Week 6 (4 hours) The subject will be asked to come to clinic before he/she takes the daily dose of study medication. The subject is asked to bring your study medications with them, and to take the study medication in the presence of the study staff, who will note the time. He/she will be asked brief medical questions and receive a physical exam and a detailed test of brain and nerve function. The subject will be asked questions about emotions, memory function, and ability to do simple tasks. The subject will have a blood test (about 2 tablespoons) to check kidney and liver function, and to check for anemia. The subject will have an EKG. If she is a woman able to become pregnant she will be asked to have a urine pregnancy test.

After the Week 6 visit is completed, and if blood and other tests indicate that the subject is still eligible, the subject will be invited to enter the Part II phase of the study. In the Part II phase,and sign a new consent. In Part II all subjects will receive ConcertaTM for the next 8 weeks. After the new consent is signed, the subject receives a two week supply of Concerta.

Week 8 (1 hour) The subject will be asked brief medical questions and receive a brief physical exam and an EKG if indicated. He/she will be given a 2 week supply of Concerta.

Week 10 (1 hour) The subject will be asked brief medical questions and receive a brief physical exam and an EKG if indicated. If she is female she will be asked to give urine for a pregnancy test .The subject will be given a new 2-week supply of Concerta.

Week 12 (1 hour) The subject will be asked brief medical questions and receive a brief physical exam and an EKG if indicated. He/she will be given a 2 week supply of Concerta.

Week 14 (4 hours) The subject will be asked brief medical questions and receive a physical exam including vital signs and a detailed test of brain and nerve function. He/she will be asked questions about emotions, memory function, and ability to do simple tasks. She/he will again receive memory questionnaires and a quality of life questionnaire. She/he will receive an EKG. If she is a woman able to become pregnant she will be asked to have a urine pregnancy test. After thisvisit the study ends.

ELIGIBILITY:
Inclusion Criteria:

Men and women 18 years of age or older and less than 65 years of age.

Able to read and understand English.

HIV infected on stable ART regimen for 5 months or greater, and not likely to change regimen for the duration of the study.

Significant dementia but able to give consent (International HIV Dementia Scale score <10).

Significant cognitive slowing on screening, defined as 1 SD below normal (t-score >60) on the Conner's CPT-II reaction time test.

Beck Depression Inventory score <16.

Documented HIV-1 RNA PCR <50 copies/mL and documented CD4 count >200 within 3 months of entry visit.

Baseline CBC and chemistry panel Grade 1 or normal.

For females of reproductive potential (women who have not been post-menopausal for at least 24 consecutive months, i.e., who have had menses within 24 months prior to study entry), or women who have not undergone surgical sterilization, specifically hysterectomy or bilateral oophorectomy or tubal ligation) will require a negative serum or urine pregnancy test within 48 hours prior to entry.

NOTE: Subject reported history is considered acceptable documentation of hysterectomy, bilateral oophorectomy, tubal ligation, tubal micro-inserts, menopause, and vasectomy/azoospermia.

All subjects must agree not to participate in the conception process (e.g., active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization), and if participating in sexual activity that could lead to pregnancy, the subject/partner must use at least two reliable methods of contraception, (condoms, without a spermicidal agent; a diaphragm or cervical cap without spermicide; an IUD; or hormone-based contraceptive), for 2 weeks before study treatment, while receiving study treatment, and for 6 weeks after receiving study treatment.

Ability and willingness of subject to provide informed consent.

Exclusion Criteria:

Inability to give informed consent. No proxy consent allowed.

Uncontrolled hypertension (SBP >140 and DBP >90 at screening and baseline).

Untreated hypogonadism, hypothyroidism or hyperthyroidism.

Initiation of antidepressants, thyroid medication or anabolic steroids within 6 weeks of screening visit.

Pregnancy or breast feeding.

Clinically significant EKG abnormalities at screening.

History of coronary artery disease, atherosclerotic disease, left ventricular hypertrophy, cardiomegaly, syncope, congestive heart failure, myocardial infarction, pacemaker, clinically significant arrhythmia, angina, history of treatment for arrhythmia.

Brain related opportunistic infections, stroke, intracranial lesions/disease, or meningitis.

History of epilepsy.

Untreated depression.

Uncontrolled diabetes (glucose <70 or >200 at screening).

Use of interferon or ribavirin during study and for 1 month prior to screening.

History of bipolar disorder, Alzheimer's dementia, ALS, Parkinson's disease or other medical dementias other than HIV-related.

History of schizophrenia, mania or other serious mental illness.

History of methylphenidate allergy.

Other serious concurrent medical illness other than HIV.

History of radiation therapy to the brain or brain injury.

History of crystal methamphetamine, cocaine, LSD use or other recreational substance use other than marijuana within the 12 months prior to screening and for the duration of the study.

Plan to use marijuana or marinol during the entire study duration and one month prior to screening visit.

Plan to drink 7 or more alcoholic drinks per week during the 4 weeks prior to screen visit and for the duration of the study.

History of alcohol dependence, alcohol abuse, cocaine addiction, crystal methamphetamine addiction or other recreational drug addiction or treatment for addiction or dependence within 5 years of screening visit.

If subject is using prescription narcotics, should be on a stable dose for at least 1 month prior to screening and throughout the study.

Previous use of Concerta™, Ritalin™, atomexitine or Adderall™ or other psychostimulants (e.g. modafinil, armodafinil) for 3 months prior to screening visit and for duration of the study.

History of tic disorders in the past 3 months or any history of Tourette's syndrome.

Greater than 10% below ideal body weight (IBW for men = 50 kg + 2.3 kg per inch over 5 feet of height, and IBW for women = 45.5 kg + 2.3 kg per inch over 5 feet of height)

Uncontrolled migraine headaches.

History of short gut syndrome, Meckel's diverticulum, or cystic fibrosis.

Family history of sudden cardiac death in a young relative.

History of fainting with exercise.

History of attention deficit disorder will be excluded, defined as a score greater than 6 on the Childhood ADHD Symptoms Scale.

-

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Change in rate of reaction time as measured by neuropsychological testing | 10 weeks of study drug exposure
  The Conner's CPT-II at screening, and at weeks 1, 5, and 14.

SECONDARY OUTCOMES:
Number of Subjects with Adverse Events as Measures of Safety and Tolerability of Concerta in HIV infected adults | 10 weeks of drug exposure
  The number of subjects who develop adverse events while on study medication vs placebo will be used to measure the safety and tolerability of ConcertaTM at 36 mg a day in this population of adult subjects with HIV over both a two week and eight week treatment period. These measures are EKG changes, electrolyte, creatinine, liver function tests, blood pressure, quality of life and sleep quality scales.

CONTACTS AND LOCATIONS:
Overall Officials: Ardis A Moe, M.D., Principal Investigator — UCLA Center for AIDS Research and Educationi
Locations (1):
- UCLA CARE Clinic, Los Angeles, California, United States